CLINICAL TRIAL: NCT05056363
Title: In The Light of Isokinetic Test and sEMG: How Effective Is Core Stability Exercise Training On Cobb Angle Muscle Strenght and Quality of Life In Adolescent Idiopathic Scoliosis
Brief Title: The Effects of Core Stability Training in Children With Adolescent Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Fuat Gokdemir, Research Assistant, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IUFGokdemir01
Record Dates: First submitted 2021-09-15; First posted 2021-09-24 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Isokinetic Testing; EMG Biofeedback; Core Stability

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): The control group will be given home based traditional scoliosis exercise training for 8 weeks, 5 days a week for 45 minutes.
  Interventions: Other: Home Based Traditional Scoliosis Exercises
- Training Group (Experimental): In addition to conventional home based traditional scoliosis exercises, patients in this group will also receive core stabilization exercise training for 45 minutes, 5 times in a week for 8 weeks. Every two sessions will be supervised in a clinic per week.
  Interventions: Other: Home Based Traditional Scoliosis Exercises; Other: Core Stability Training

INTERVENTIONS:
Other: Home Based Traditional Scoliosis Exercises — Patients in this group will receive posture exercises, strengthening exercises, diaphragmatic breathing exercises and stretching exercises.
Other: Core Stability Training — Patients in this group will receive traditional scoliosis exercises. In addition, the training group will receive core stabilization exercises for multifidus, diaphragm,erector spines, rectus abdominis, internal and external obliques, quadratus lumborum, iliopsoas, gluteus maximus, and pelvic floor muscles.
  Arms: Training Group

SUMMARY:
Adolescent idiopathic scoliosis (AIS) is a three-dimensional structural deformity of the spine in which lateral flexion and axial rotation are seen in vertebrae with a Cobb (method for measuring spinal curvature) angle of 10° and above. AIS is the most common type of scoliosis and it occurs in the period from the onset of puberty (up to 10 years) until the closure of growth plates.

Children with AIS have cosmetic effects, decrease in functional capacity, muscle weakness in certain parts of the body, decrease in quality of life and posture disorders. Lack of core stability might be causing these problems.

Core stability training may have a positive effect for these problems experienced by children with AIS.

Pathologies that cause the disease may originate from the nervous system and musculoskeletal system. In this study, the investigators will evaluate these systems objectively with EMG biofeedback and Isokinetic Testing.

The aim of this study is to show the effect of core stability training on various problems (as we mentioned before) caused by the disease. In addition, the investigators of this study hope to contribute to the literature(with objective evaluations) about the pathological background and treatment of this challenging disease which the cause is unknown.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with AIS between the ages of 10-20
* Cobb angle is between 15-40 degrees
* The child's and family's consent to participate in the study
* The child does not receive any other treatment that will affect his scoliosis.

Exclusion Criteria:

* Surgical operation in the last 3 months
* Presence of an orthopedic, neurological, systemic disease that will prevent him from exercising
* Having mental, communicative and behavioral disorders that may cause problems understanding commands and questions or performing exercises
* Exercising 3 or more days a week.

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Muscle Strength of Trunk Flexion / Extension | 8 week
  Measurement of isokinetic and isometric muscle strength with Biodex System 3Pro Multijoint System Isokinetic Dynamometer.
Cobb Angle | 8 week
  Cobb Angle measurement with AP Radiography
Muscle Strength | 8 week
  Evaluation of the muscle strength with using a non-invasive Myomed 932 EMG-biofeedback device (Enraf-Nonius, The Netherlands)
Muscle Electromyographic Activity | 8 week
  Measurement of the surface electromyographic activity with using a non-invasive Myomed 932 EMG-biofeedback device (Enraf-Nonius, The Netherlands)

SECONDARY OUTCOMES:
Trunk Rotation | 8 week
  Evaluation of the thoracic, thoracic-lumber junction, lumber axial trunk rotation with Bunnell Scoliometer
Patients Quality of Life | 8 week
  Quality of life will be measured with using the Scoliosis Research Society 22 item questionnaire (SRS-22r).
  SRS-22 has a minimum score of 22 and a maximum score of 110. Each question is scored on 1-5 scale. Questions are sorted into different domains and total and mean scores for each domain are calculated. A total score for the entire questionnaire is also calculated.
Cosmetic Deformity Evaluation | 8 week
  Patients cosmetic deformity will be evaluated with Walter Reed Visuel Assesment Scale.
  This scale includes seven items with figures representing different aspects of the spinal deformity: spinal deformity, rib prominence, lumbar prominence, thoracic deformity, trunk imbalance, shoulder asymmetry and scapular asymmetry. The figures are scored from minimum (1, no deformity) to maximum (5, severe deformity) and summed up to yield a total score (minimum: 5 points, maximum: 35 points).
Flexibility Measurement | 8 week
  Patients flexibility will be measured with forward and lateral bending tests

CONTACTS AND LOCATIONS:
Overall Officials: Fuat Gökdemir, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided